CLINICAL TRIAL: NCT00965809
Title: Double Blind, Placebo-Controlled Trial of THC as add-on Therapy for PTSD
Brief Title: Add on Study on Δ9-THC Treatment for Posttraumatic Stress Disorders (PTSD)
Acronym: THC_PTSD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arieh Y. Shalev, M.D. / Head, Department of Psychiatry, Hadassah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THC09
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-09

CONDITIONS: Posttraumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- ACTIVE THC (Experimental): Subjects will take 5MG of THC in 6 drops of olive oil orally.
  Interventions: Drug: Tetrahydrocannabinol
- Placebo (Placebo Comparator): Subjects will take 6 drops of olive oil orally twice a day from an identical vial than those in the active arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tetrahydrocannabinol — Five mg. of THC in 6 drops of olive oil orally twice a day for 6 weeks.
  Arms: ACTIVE THC
Other: Placebo — Subjects will take 6 drops of olive oil orally twice a day from an identical vial than those in the active arm
  Arms: Placebo

SUMMARY:
Stress Disorder (PTSD) is a chronic and debilitating anxiety disorder which is widespread in every social level and is very prevalent in outpatient and inpatient settings.

A recent open-label study showed that the synthetic cannabinoid receptor agonist Nabilone had beneficial effects abolishing or greatly reducing nightmares that persisted in spite of treatment with conventional PTSD medications. Furthermore, a big number of patients suffering from chronic PTSD report using smoked marijuana because its tranquilizing effect and sleep quality improvement. According to clinical and epidemiological data different derivates from the cannabis plant are illegally and pervasively consumed by PTSD patients in order to reduce distress.

The aim of the proposed study is to broaden the previous observations and to measure the extent to which Δ 9-THC will bring to significant improvement on the full spectrum of PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between the 19-60 years of age with a diagnosis of PTSD.
* Women must not be currently pregnant and must use a reliable method of contraception for the duration of the study.
* Subjects must be on stable medication (4 weeks minimum) for their PTSD (symptomatic despite current treatment), must be able to provide written informed consent, must be able adequately understand and comply with the study's instructions and protocol .

Exclusion Criteria:

* Those not meeting the inclusion criteria and those not able to give informed consent.
* Women who are currently pregnant or nursing.
* Those at immediate risk of harming self or others; those who have a clinically significant medical illness or other significant psychiatric illness;
* currently abusing alcohol or drugs;
* currently being treated with an investigational medication or medication that is contraindicated with cannabinoids;
* have a known allergy to cannabis-based products.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale | Baseline and end o ftreatment

SECONDARY OUTCOMES:
Nightmare Frequency Questionaire Score | Baseline Weeks 3 &6 (EOS)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel